CLINICAL TRIAL: NCT04584008
Title: A Real-world Study to Explore and Evaluate Individualized Targeted Agents for Patients of Digestive Cancers Based on Molecular Characteristics After Standard Therapy Failure in China
Brief Title: Targeted Agent Evaluation in Digestive Cancers in China Based on Molecular Characteristics
Acronym: VISIONARY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Hangzhou DIAN Medical Diagnostic Center Co., Ltd., China (Unknown); 3D Medicines (Industry)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGS01
Record Dates: First submitted 2020-09-21; First posted 2020-10-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Biliary Tract Neoplasms; Gastric Cancer; Esophageal Squamous Cell Carcinoma; Colorectal Cancer; Gastrointestinal Stromal Tumors; Pancreatic Cancer; Neuroendocrine Tumors; Unknown Primary Cancer; Digestive Cancer
Keywords: Umbrella Study; Next Generation Sequence
MeSH Terms: conditions — Biliary Tract Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma; Colorectal Neoplasms; Gastrointestinal Stromal Tumors; Pancreatic Neoplasms; Neuroendocrine Tumors; Neoplasms, Unknown Primary; Gastrointestinal Neoplasms | interventions — Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Matched Targeted Agent (Experimental): Matched Targeted Agent
  Interventions: Drug: FGFR Inhibitor, IDH1 Inhibitor, HER2 Inhibitor, PARP Inhibitor, BRAF Inhibitor, MEK Inhibitor, ICIs, EGFR-TKIs, NTRK-TKI, and et. al.
- Unmatched Therapy (Active Comparator): Unmatched Therapy
  Interventions: Drug: Other Therapy

INTERVENTIONS:
Drug: FGFR Inhibitor, IDH1 Inhibitor, HER2 Inhibitor, PARP Inhibitor, BRAF Inhibitor, MEK Inhibitor, ICIs, EGFR-TKIs, NTRK-TKI, and et. al. — According to the treatment dose approved by NMPA/FDA, evaluation will be conducted every 2 cycles until tumor progression or adverse events cannot be tolerated.
  Other Names: Targeted Agent
  Arms: Matched Targeted Agent
Drug: Other Therapy — Patients will receive other treatments, including cytotoxic drugs, antiangiogenic drugs, best supportive care, clinical trials of unmatched new drugs, etc..
  Other Names: Other Drugs
  Arms: Unmatched Therapy

SUMMARY:
This a prospective real-world navigation study using tumor DNA sequencing technology to sequence genes of previously treated and refractory gastrointestinal tumors, which are generally considered to be highly heterogeneous and complex, to screen potential molecular targeted drugs for individualized treatment. This study may provide feasibility and response information, which will be the basis for designing better randomized trials, which may change the pattern of cancer treatment. If the hypothesis is finally proved, it will help doctors and molecular biologists to choose the best drug (or combination of drugs) based on the individual oncogenomics of each patient.

DETAILED DESCRIPTION:
This is a prospective, open label, real-world study to evaluate the feasibility of matched molecular targeted therapy in patients with refractory gastrointestinal cancer based on tumor molecular characteristics as standard treatment failure. This is a non-randomized trial designed to test molecular matching strategies based on patient genome information. The molecular tumor board (MTB) will recommend treatment, but the treatment decision is up to the attending physician. FoundationOne CDx was used for tissue genomic analysis. If possible, PD-L1 immunohistochemistry (IHC), tumor mutation load (TMB), and microsatellite instability (MSI) status will also be evaluated. Based on this information, MTB, composed of multidisciplinary experts, will focus on the selection of customized, best matched drugs or combinations to target most of the genomic changes in each patient, also taking into account potential drug toxicity. The final treatment will be based on the choice of oncologists, who will formulate treatment plan by combining MTB discussion, patient preference, attention to complications, consideration of drug toxicity, insurance coverage of off label drugs and availability of clinical trials of research drugs, thus reflecting the actual clinical practice nowadays in China. The acquisition of drugs follows the actual situation in the real world and is not within the scope of this study design.

The principles of MTB treatment recommendations can be referred to the NCI-MATCH trial:

Grade 1: FDA / NMPA approval; clear evidence and mechanism; concomitant diagnostic relationship between drug and target.

Grade 2: The drug reaches the clinical end point (objective response rate, PFS or OS); there is evidence of target inhibition; there is strong evidence to predict relationship between the target and the drug.

Grade 3: The drug has evidence of clinical activity and target inhibition; there is some evidence to predict the relationship between target and drug.

Grade 4: Pre-clinical evidence of anti-tumor activity and evidence of target inhibition; there is hypothesis to predict the relationship between target and drug.

Patients who meet the inclusion criteria and sign informed consent will be analyzed for tumor mutation by FoundationOne CDx detection. Biopsy specimens of metastatic foci can be selected for gene detection. If there is no targeted therapy among patients, the archived diagnostic tumor samples can also be used for detection. If the patient has received targeted therapy, the investigators will try to obtain biopsy samples after treatment. If the sample cannot be tested or the test results are not satisfactory, additional slices need to be sent to the laboratory. If the repeated test fails, repeat biopsy if the clinical conditions permit, or patients should be included in the unmatched treatment group.

Determining the interventability of gene mutations depends on genomic changes, allele frequency, and diagnosis. This study will combine the recommendations of MTB and gene testing reports to determine the interventability of mutated genes.

Interventional mutation: cancers have FDA or NMPA approved therapies, or there are matching drugs in clinical trials.

Non-interventional mutation: there is no FDA or NMPA approved treatment for cancers, and no matching drug is available in clinical trials.

MTB should at least be composed of attending doctors, molecular pathology experts and bioinformatics experts. The research center is responsible for the establishment and holding of MTB. As management of patients enrolled in this study is essential, the research committee, including but not limited to the main investigator of the study and the treated medical oncologist, can provide advice as needed between MTB meetings to avoid treatment delays. By analyzing the genomic variation of patients, independent MTB recommends molecular targeted therapy that can inhibit the mutation directly or through related pathways or be included in relevant clinical trials. The independent research committee will use the "N-to-1" model of precision medicine to propose a matching therapy consisting of at least one drug that targets molecular changes. The investigators expect 50-70% of patients to carry intervening variants, and that proportion is rising rapidly as learning more about these pathways and drugs. The investigators expect that about 40% of patients with intervening variants will be able to receive molecular targeted "matching" therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or metastatic malignant tumors of digestive tract, including but not limited to:

  1. Biliary tract cancer (including gallbladder cancer and cholangiocarcinoma)
  2. Gastric cancer
  3. Esophageal squamous cell carcinoma
  4. Colorectal cancer
  5. Gastrointestinal stromal tumor
  6. Pancreatic cancer
  7. Primary unknown metastatic carcinoma of digestive system
* failure of conventional treatment;
* have at least one measurable lesion according to RESIST1.1;
* the target lesion is not suitable for local treatment;
* the expected survival time was more than 3 months;
* age ≥ 18 years old;
* the main organs function well;
* be able to swallow and retain oral medication if necessary;
* patients must have enough tissue samples for gene mutation detection;
* informed consent signed.

Exclusion Criteria:

* main lesions were suitable for local treatment;
* serious or uncontrolled medical diseases that researchers consider to be confusing in the treatment response analysis (i.e. uncontrolled diabetes, chronic kidney disease, chronic lung disease or uncontrolled active infection, mental illness / social status that limits compliance with research requirements);
* pregnant or lactating patients or any fertile patients taking no appropriate pregnancy prevention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of patients receiving targeted agent | up to 2 years
  Objective response rate (ORR) per RECIST 1.1 criteria according to investigators assessment

SECONDARY OUTCOMES:
Proportion of patients with intervening genomic variation | up to 2 years
  Proportion of patients with intervening genomic variation
Progression Free Survival (PFS) of patients receiving targeted agent | up to 2 years
  Progression Free Survival (PFS) per RECIST 1.1 criteria according to investigators assessment
Overall Survival (OS) of patients receiving targeted agent | up to 2 years
  Overall Survival (OS) per RECIST 1.1 criteria according to investigators assessment
Number of participants with treatment-related adverse events | up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Differences of OS between 2 groups | up to 2 years
  Differences of OS between 2 groups per RECIST 1.1 criteria according to investigators assessment

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China